CLINICAL TRIAL: NCT05634642
Title: Analysis of the Inner Diameter of the Distal Radial Artery and the Influencing Factors in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Wujin People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WJH20221122
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Distal Radial Artery
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Using ultrasound to measure the diameter of distal radial artery

SUMMARY:
Cardiovascular intervention via distal radial artery (DRA) approach has become more and more extensive. However, the DRA is smaller than conventional radial artery (CRA). Assessing the size of the DRA before vascular intervention is extremely important to select suitable patients. There are still few large-sample studies to evaluate the size of DRA and its influencing factors in the Chinese population.

DETAILED DESCRIPTION:
In recent years, the clinical application of distal radial artery (DRA) approach in cardiovascular intervention has become more and more extensive. However, compared with CRA, the DRA is smaller, resulting in an increased proportion of patients requiring multiple punctures and a lower success rate of implantation. It has been found that the mismatch between artery sheath and vessel size is one of the independent risk factors for postoperative vascular approach complications. Therefore, assessing the size of the DRA before vascular intervention is extremely important to select suitable patients, improve the success rate of puncture, and reduce the complications associated with the approach There are still few large-sample studies to evaluate the size of DRA and its influencing factors in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is prepare for coronary angiography

Exclusion Criteria:

* Lack of upper limbs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who is prepare for coronary angiography
Sampling Method: Probability Sample
Enrollment: 1182 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Diameter of distal radial artery | 24 hours before coronary intervention
  Measure the diameter of distal radial artery in anatomic snuffbox by ultrasound

SECONDARY OUTCOMES:
Diameter of conventional radial artery | 24 hours before coronary intervention
  Measure the diameter of conventional radial artery by ultrasound
Diameter of ulnar artery | 24 hours before coronary intervention
  Measure the diameter of ulnar artery by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Cai, Dr., Study Chair — Wujin hospital affiliated with Jiangsu University
Locations (1):
- Changzhou Wujin People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Result] Li F, Shi GW, Yu XL, Song RX, Xiao JQ, Huang HM, Li LM, Zhang LY, Gong C, Cai GJ. Safety and efficacy of coronary angiography and percutaneous coronary intervention via distal transradial artery access in the anatomical snuffbox: a single-centre prospective cohort study using a propensity score method. BMC Cardiovasc Disord. 2022 Mar 2;22(1):74. doi: 10.1186/s12872-022-02518-8. PMID 35236288
- [Result] Eid-Lidt G, Rivera Rodriguez A, Jimenez Castellanos J, Farjat Pasos JI, Estrada Lopez KE, Gaspar J. Distal Radial Artery Approach to Prevent Radial Artery Occlusion Trial. JACC Cardiovasc Interv. 2021 Feb 22;14(4):378-385. doi: 10.1016/j.jcin.2020.10.013. PMID 33602433
- [Result] Norimatsu K, Kusumoto T, Yoshimoto K, Tsukamoto M, Kuwano T, Nishikawa H, Matsumura T, Miura SI. Importance of measurement of the diameter of the distal radial artery in a distal radial approach from the anatomical snuffbox before coronary catheterization. Heart Vessels. 2019 Oct;34(10):1615-1620. doi: 10.1007/s00380-019-01404-2. Epub 2019 Apr 10. PMID 30972548
- [Result] Naito T, Sawaoka T, Sasaki K, Iida K, Sakuraba S, Yokohama K, Sato H, Soma M, Okamura E, Harada T, Yoshimachi F. Evaluation of the diameter of the distal radial artery at the anatomical snuff box using ultrasound in Japanese patients. Cardiovasc Interv Ther. 2019 Oct;34(4):312-316. doi: 10.1007/s12928-018-00567-5. Epub 2019 Jan 7. PMID 30617776